CLINICAL TRIAL: NCT02044705
Title: Impact of Active and Healthy Families (Familias Activas y Saludables): A Family-Based Group Medical Appointment Model for Childhood Obesity in Federally Qualified Health Centers
Brief Title: Impact of Active and Healthy Families
Acronym: AHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-07-4508 A; 033728 (Other Grant/Funding Number: Safeway Foundation)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Overweight; Obesity
Keywords: Primary Health Care; Pediatrics; Obesity; Overweight; Clinical trial; Hispanic Americans; Family; Body mass index
MeSH Terms: conditions — Overweight; Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family group sessions (Experimental): Active and Healthy Families
  Interventions: Behavioral: Active and Healthy Families
- Wait-list control (No Intervention): Controls may participate in Active and Healthy Families after the study

INTERVENTIONS:
Behavioral: Active and Healthy Families — Pediatric obesity intervention delivered through five bi-weekly Active and Healthy Families family-based group medical appointments (i.e., sessions).
  Arms: Family group sessions

SUMMARY:
The purpose of this study is to evaluate the impact of the 10-week Active and Healthy Families (AHF) intervention on body mass index (BMI) in Latino youth aged 5-12 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5-12 years
* Body mass index greater than or equal to the 85th percentile for age and sex
* Patients seen at Contra Costa County clinics participating in Active and Healthy Families
* Spanish speaking
* Parent of participant

Exclusion Criteria:

* Previous participation in Active and Healthy Families

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in body mass index (BMI) | Baseline and at week 10
  Change from baseline are assessed from measured height and weight

SECONDARY OUTCOMES:
Change from baseline in blood glucose | Baseline and week 10
Changes from baseline in fasting lipids | Baseline and week 10
Change from baseline in insulin resistance | Baseline and week 10
Change from baseline in blood pressure | Baseline and week 10

OTHER OUTCOMES:
Change in parent weight | Baseline and week 10

CONTACTS AND LOCATIONS:
Overall Officials: Kristine A Madsen, MD, Principal Investigator — University of California, Berkeley
Locations (2):
- United States (2):
  - Pittsburg Health Center, Pittsburg, California
  - West County Health Center, San Pablo, California